CLINICAL TRIAL: NCT02877511
Title: Supervised Outdoor-Use Test For Sunscreen Products in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 18803
Record Dates: First submitted 2016-08-19; First posted 2016-08-24 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): 2/3 of subjects testing the test article
  Interventions: Drug: BAY987517
- Arm 2 (Active Comparator): 1/3 of subjects testing the marketed control
  Interventions: Drug: Sunscreen Lotion (Y65-110)

INTERVENTIONS:
Drug: BAY987517 — Applied liberally to the skin (Formulation: Y73-161
  Arms: Arm 1
Drug: Sunscreen Lotion (Y65-110) — Applied liberally to the skin
  Arms: Arm 2

SUMMARY:
To assess the safety of a sunscreen product under supervised outdoor-use conditions

ELIGIBILITY:
Inclusion Criteria:

* Subject must be healthy, males or females between 18 to 65 years of age with no medical conditions of the skin.
* Subjects must have Fitzpatrick Skin Type I, II, III or IV.
* Subjects must agree to restrict their sun exposure activities for at least five days immediately preceding participation in the study.

Exclusion Criteria:

* Subjects must not have actinic keratoses, skin cancer, psoriasis, eczema, or any other acute or chronic skin conditions.
* Subjects must not have visible erythema, blistering, or peeling that would indicate recent sunburn as determined by the baseline skin evaluation.
* Subjects must not have significantly tanned skin.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2016-08-20 (Actual); Primary Completion 2016-08-21 (Actual); Study Completion 2016-08-21 (Actual)

PRIMARY OUTCOMES:
Skin response to sun exposure according to the Skin Evaluation Response Scale from 0 to 3 | From the beginning of the study until 24 hours after study

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States